CLINICAL TRIAL: NCT07092852
Title: Pharmacogenomic-Based Medication Safety Reviews of Persons With Intellectual and Developmental Disabilities
Brief Title: PGx Medication Safety Reviews of Persons With IDD
Status: Not yet recruiting | Type: Observational
Sponsor: GalenusRx, Inc. (Industry)
Collaborators: CP Unlimited (Unknown)
Responsible Party: Sponsor
Other Study IDs: GRx-PGx001_CPU_2025
Record Dates: First submitted 2025-07-08; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Intellectual Disability, Mild; Intellectual Disability, Mild to Moderate; Developmental Disability
Keywords: Intellectual disabilities; Developmental disabilities; IDD; pharmacogenomics
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residents of CP Unlimited: All persons residing in CPU facilities during the study period will be included in the study, except those who are under 21 years of age, in whom a cheek swab cannot be obtained, and those who for whom no valid consent for participation is in place.
  Interventions: Other: Cheek swab for PGx testing; Other: Medication safety review

INTERVENTIONS:
Other: Cheek swab for PGx testing — Pharmacogenetic test kits will be provided to each CPU residence. An order will be issued to obtain samples for the study - a cheek swab - to be collected by residence direct care providers or nursing staff, trained in the procedure for obtaining the sample, and preparing and submitting it for transport. Failures to collect and submit valid samples, the number of samples submitted that cannot be processed, and the reasons for failure, will be recorded. If a submitted sample cannot be processed, another sample can be obtained and submitted.
Other: Medication safety review — A medication reconciliation will be performed by a GalenusRx pharmacist on all included residents. Medication data for enrolled participants will be collected by the GalenusRx pharmacist from the unique pharmacy provider and/or the medication records from the facility and a medication reconciliation will be conducted with the nurse of the residents' facility. GalenusRx pharmacists will apply a CDSS to patients' medication regimens, screening for drug interactions, assess medication related risks, and consider pharmacogenomic type and phenoconversion results in recommending appropriate drug selection and dosage to prescribing clinicians.

SUMMARY:
The purpose of this study is to assess the feasibility of a comprehensive medication review and PGx initiative as part of the care process for individuals in the care of CP Unlimited. This initiative may help improve management of medications and overall health and well-being for participating individuals. Please note that in the context of the research being conducted, all information will remain confidential and deidentified for analyses.

Under the proposed study protocol, CP Unlimited, in partnership with pharmacists at GalenusRx, will implement and assess a comprehensive medication safety and PGx initiative. Almost three quarters of all clinical trials have eligibility criteria resulting in the exclusion of adults with IDD. This study will help address ongoing health practice disparity. As indicated above, the investigators are requesting the authorization of the guardian or representative, on behalf of the participant under their supervision, to enroll this individual in the proposed study because she/he is currently prescribed medications or may eventually receive prescribed or over-the-counter medications. Hereinafter, the denomination "he/she, him/her, his/her or them/their" will be used to refer to the individual with IDD.

The response to medication can be affected by variations in our genes and by other medications and various disease conditions. Information contained in our genes can vary from one patient to another patient and this can explain why we all can respond differently to medications. Genetic testing and a review of his/her medications can help to determine if the medication will work for him/her. PGx is how his/her genes affect the way he/she responds to specific drugs. PGx can tell if he/she is more or less likely to feel bad reactions to a drug, or if a drug is likely to benefit him/her and be safe for him/her to take. Knowing his/her genetic information and all medicines that he/she is taking can help his/her pharmacist and his/her doctor find the combination of medicines that will work the best for him/her, now and in the future.

DETAILED DESCRIPTION:
The impact of polypharmacy, defined as the use of five or more medications daily, to manage multiple conditions is well recognized in general and elderly populations (1,2), and in persons with intellectual and developmental disabilities [IDD] (3,4). People with IDD are living longer than in the past. However, individuals with IDD have more chronic conditions that require medications for treatment than the general population and often receive care and medications from several clinicians (5-9).

The use of multiple medications is associated with an increased risk of adverse drug events [ADEs] and is a significant cause of morbidity and death (10). Annually, adverse drug events (ADEs) in outpatient settings lead to an estimated one million emergency department visits and roughly 125,000 hospital admissions (11). Pharmacogenomic (PGx) testing-a tool that can be utilized to identify genetic variants known to impact drug response-has the potential to inform, reduce and prevent ADEs (12). GalenusRx's investigators have conducted research, developed programs and products over the last 25 years, and demonstrated that pharmacists' interventions can prevent ADEs, decrease hospitalizations, emergency department visits, falls, hospital readmission and even premature mortality (13,14, 15).

Constructive Partnerships Unlimited [CPU] serves people with cerebral palsy and other IDD, and their families, in New York City and surrounding communities, with day programs and residential programs that are the focus of this proposal. CP Unlimited was created by groups of parents of disabled children from around New York State when, in 1946, they formed an association to increase public awareness, sponsor parent and professional training, encourage research, and engage in legislative advocacy for the development of services needed for their children. By 2018, CP of New York State had evolved into a broad-based, multi-service organization serving persons with all types of IDD. In June of that year, the Agency established its Hudson Valley Division to provide residential, day habilitation, and Article 16 clinical services to adults with IDD throughout Putnam and Dutchess Counties. The organization now includes Metro Services and Metro Community Health Centers located in New York City, an Affiliate Services office in Albany, New York, and twenty-four Affiliates throughout New York State. In 2019, the organization shifted its focus to the New York City and beyond to better care for a growing population of people with IDD in need of support. Their suite of options featured enhanced community living, day programs, vocational and employment programs, medical and clinical services, early intervention, educational, recreational, and family support services. Currently, more than 700 people are in CPU residential programs and are served by a single pharmacy, TotalCareRx, for drug dispensing.

GalenusRx is an advanced clinical pharmacy technology and consulting service and non-dispensing pharmacist company. It collaborates with prescribers and dispensing pharmacies to optimize drug regimen's outcomes and avoid ADEs. GalenusRx goal is to reduce predictable and preventable medication-related problems and ADEs. GalenusRx pharmacists provide personalized evidence-based PGx consults and PGx focused medication safety reviews. GalenusRx personalized pharmacy services are aided by a proprietary, evidence-based clinical decision support system (CDSS) APPRAISETM (Actionable PolyPharmacy Risk Assessment Index for Safety and Equity) that supports pharmacists with the identification of drug-drug interactions, drug-gene interactions and drug-drug-gene interactions. Based on the clinical pharmacist's interpretation and professional judgement, subsequent actionable recommendations are provided and/or discussed with the health care providers (e.g., for dose adjustments, alternative agent selection, monitoring therapy response, ADE monitoring).

CP Unlimited organization in partnership with GalenusRx proposes to conduct a study to assess the feasibility of medication safety reviews and pharmacogenomics as part of a consolidative care process for individuals with IDD.

Achieving a therapeutic response to a drug often requires balancing desired drug effects and undesired side effects. To find the right drug, and the right dose for the right patient often requires titration of the dose, depending on the individual patient's response to the drug. Patients' responses are influenced by many factors, including their body size, kidney or liver function, environment, concomitant illnesses, and other substances they are exposed to, including tobacco or alcohol, and other drugs, among others.

Individual patients' genetic make-up is known to affect their responses to drugs. Individuals may have a genetic predisposition to eliminate drugs [or convert them to another form that may be more active, less active or inactive] at faster or slower rates than others do. Knowledge of individual patient's genetic make-up, so far as it influences their response to drugs, is not as widely known or available as other factors that may influence their response to drugs. Availability of information of individuals' genetic make-up affecting drug handling has potential to improve medication safety.

Patients with IDD are more frequently than the general population prescribed drugs with narrow therapeutic indices ['safety margins,' in common language] and drugs prone to interact with other drugs. Among these are many psychotropic or psychiatric medications, and antiseizure medications. Also, ADEs and drug-interactions may be more difficult to detect, due to patients' limitations on expressing themselves; consequently, ADEs may be exacerbated in IDD patients, because of concomitant diseases or limitations.

Knowledge of a patient's pharmacogenomic status has the potential to guide medication management and utilization, hence improving treatment safety and efficacy. The potential for such improvement is of particular importance in IDD populations. Most clinical trials have eligibility criteria leading to exclusion of certain groups, particularly adults with IDD, due to the complexity of their medical conditions and drug regimens. Integration of PGx testing and results remains very limited in clinical practice for vulnerable population, including adults with IDD.

This prospective observational study to assesses the feasibility of integrating pharmacogenomic-based medication regimen safety reviews, as part of a comprehensive care process, addressing polypharmacy issues in a population of persons with intellectual and developmental disabilities (IDD).

ELIGIBILITY:
Inclusion Criteria:

* Beneficiary with IDD
* Reside in a CP Unlimited facility, NY state
* At least 21 years of age

Exclusion Criteria:

* Pregnant
* Medical or physical abnormality that prevents cheek swab collection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons residing in CPU facilities during the study period will be included in the study, except those who are under 21 years of age, in whom a cheek swab cannot be obtained, and those who for whom no valid consent for participation is in place. Beneficiaries will be identified by the CMO and/or the medical care team of the project. The number of persons excluded and the reasons for exclusion will be reported and analyzed. All residents have current consent for standard medical care, subject to individual 'carve-outs.' Any procedures or analyses performed on any individual in the course of this research project.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Measure the Feasibility of PGx Testing in IDD Population | Two years
  Measure feasibility of a PGx testing program calculating the number of pharmacogenetic tests / medication safety reviews completed.
Measure the Acceptability of Implementing a PGx Program | Two years
  Measure the acceptability of implementing a PGx program by examining the recommendations accepted and transferred to a dispensing pharmacy.

SECONDARY OUTCOMES:
Identify the PGx Profile of CP Unlimited Patients | Two years
  The PGx profile of CP Unlimited patients will be measured by quantifying the frequencies of which genes in drug-gene interactions are observed.
Identify Drug and Drug Classes of Drug-Gene and Drug-Drug-Gene Interactions | Two years
  Drug and drug classes will be identified by quantifying the frequency in which drug-gene and drug-drug-gene interactions are associated with recommendations.
Program Feasibility Considering Data Collection | Two years
  Program feasibility will be measured by the examining the ratio of cheek swabs completed to the the percentage of samples requiring a second review.

OTHER OUTCOMES:
Personalized Medication Safety Management, Genetic Results, and Acceptance | Two years
  To explore the relationship between PMSM, genetic results and acceptance using an investigator developed clinician satisfaction survey. Likert scales will be used, where the higher score indicates higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, BPharm, MSc, PhD, Principal Investigator — GalenusRx, Inc.; Ira Salom, MD, Principal Investigator — CP Unlimited
Locations (2):
- United States (2):
  - GalenusRx, Inc., Montverde, Florida
  - CP Unlimited, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the context of this study. Data may be published, but will be deidentified or of the whole study population.

REFERENCES:
- [Background] Holden B, Gitlesen JP. Psychotropic medication in adults with mental retardation: prevalence, and prescription practices. Res Dev Disabil. 2004 Nov-Dec;25(6):509-21. doi: 10.1016/j.ridd.2004.03.004. PMID 15541629
- [Background] Doan TN, Lennox NG, Taylor-Gomez M, Ware RS. Medication use among Australian adults with intellectual disability in primary healthcare settings: a cross-sectional study. J Intellect Dev Disabil. 2013 Jun;38(2):177-81. doi: 10.3109/13668250.2013.778968. Epub 2013 Apr 3. PMID 23550741
- [Background] Aman MG, Lam KS, Van Bourgondien ME. Medication patterns in patients with autism: temporal, regional, and demographic influences. J Child Adolesc Psychopharmacol. 2005 Feb;15(1):116-26. doi: 10.1089/cap.2005.15.116. PMID 15741793